CLINICAL TRIAL: NCT01192802
Title: Effect of Intestinal Helminths on Gut Microflora
Brief Title: Efficacy of Albendazole to Treat Intestinal Helminths and Its Effect on Gut Microflora
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Responsible Party: Dr Ayola Akim ADEGNIKA, Medical Research Unit
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Albendazole-001
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Intestinal Diseases; Helminthiasis
Keywords: albendazole; ascaris; trichiurus; hookworms
MeSH Terms: conditions — Intestinal Diseases; Helminthiasis; Hookworm Infections | interventions — Albendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 dose, Albendazole , tablet (Active Comparator)
  Interventions: Drug: albendazole
- 2 doses, albendazole, tablet (Active Comparator): 1 tablet of 400 mg of albendazole per day for two consecutive days
  Interventions: Drug: albendazole
- 3 doses albendazole, 400mg, tablet (Active Comparator)
  Interventions: Drug: albendazole

INTERVENTIONS:
Drug: albendazole — 1 tablet of 400 mg of albendazole per day for three consecutive days
  Arms: 3 doses albendazole, 400mg, tablet
Drug: albendazole — single 1 tablet of 400 mg of albendazole
  Arms: 1 dose, Albendazole , tablet
Drug: albendazole — 1 tablet of 400 mg of albendazole per day for two consecutive days
  Arms: 2 doses, albendazole, tablet

SUMMARY:
Albendazole is a main anti-helminth, however there is a lack of data regarding its efficacy in the school children population. The aim of this study is to evaluate the efficacy of the albendazole one versus two and three doses, in school children infected with intestinal helminth.

ELIGIBILITY:
Inclusion Criteria:

* presence of intestinal helminths eggs in the stool

Exclusion Criteria:

* allergy to imidazole derivate
* No intestinal helminths

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
parasite cleared and reduced up to 80% at day 42 | 42 days

SECONDARY OUTCOMES:
Prevalence of major gut bacteria | 42 days
  Change in the prevalence of major gut bacteria after antihelminth treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical research Unit of Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Derived] Adegnika AA, Zinsou JF, Issifou S, Ateba-Ngoa U, Kassa RF, Feugap EN, Honkpehedji YJ, Dejon Agobe JC, Kenguele HM, Massinga-Loembe M, Agnandji ST, Mordmuller B, Ramharter M, Yazdanbakhsh M, Kremsner PG, Lell B. Randomized, controlled, assessor-blind clinical trial to assess the efficacy of single- versus repeated-dose albendazole to treat ascaris lumbricoides, trichuris trichiura, and hookworm infection. Antimicrob Agents Chemother. 2014 May;58(5):2535-40. doi: 10.1128/AAC.01317-13. Epub 2014 Feb 18. PMID 24550339
- See also: Medical Research Unit of the Albert Schweitzer Hospital — http://www.lambarene.org